CLINICAL TRIAL: NCT05937191
Title: Leflunomide is Safe and Effective for the Induction and Maintenance of Idiopathic Pulmonary Hemosiderosis Remission
Brief Title: Leflunomide for Idiopathic Pulmonary Hemosiderosis in Children
Acronym: Lef for IPH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Weiping Tan, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-001
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Pulmonary Hemosiderosis; Leflunomide
Keywords: Idiopathic pulmonary hemosiderosis; Leflunomide; glucocorticoid
MeSH Terms: conditions — Hemosiderosis, Pulmonary | interventions — Leflunomide

STUDY DESIGN:
Intervention Model Description: Leflunomide+Stroid treatment Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPH Patients (Experimental): Leflunomide+Steroid treatment
  Interventions: Drug: Leflunomide
- Control Group (Active Comparator): Steroid treatment
  Interventions: Drug: Steroid Drug

INTERVENTIONS:
Drug: Leflunomide — Leflunomide+Glucocorticoids treatment Group
  Arms: IPH Patients
Drug: Steroid Drug — Steroid Treatment
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to compare Leflunomide in Idiopathic pulmonary hemosiderosis. The main questions it aims to answer are:

* The efficacy and safety of Leflunomide in Idiopathic pulmonary hemosiderosis
* The mechanism of leflunomide in treating Idiopathic pulmonary hemosiderosis Participants will be treated with leflunomide plus stroid. A comparison group: Researchers will compare the control group treated with stroid to see if the efficacy of Leflunomide would be better than control group.

DETAILED DESCRIPTION:
This study conducted a prospective, open, parallel controlled, single center clinical trial on the combination of Leflunomide and Stroid therapy for children with IPH, and conducted a one-year follow-up. The main indicators (pulmonary hemorrhage/hemoptysis frequency) and secondary indicators (serum iron metabolism level, T lymphocyte subpopulation, lung function, inflammatory cells, and inflammatory factors) were evaluated before and after treatment, Exploring the safety and effectiveness of leflunomide in the treatment of IPH, it is expected that the combination of leflunomide and conventional treatment can improve the remission rate of clinical symptoms in children with IPH, inhibit the progressive deterioration of lung function, and the research results are expected to bring new treatment methods and strategies for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 6 months to 18 years old;
2. Diagnose as IPH;
3. Parents or guardians agree to treatment and sign a written informed consent form.

Exclusion Criteria:

1. Individuals who are allergic to any ingredients used in leflunomide tablets;
2. Complicated with serious basic diseases (such as systemic malignant diseases, heart failure, liver and kidney failure, immune deficiency, serious infectious diseases, Lung transplantation or other patients with immediate surgical indications);
3. Patients with other lung diseases;
4. Have a history of abnormal coagulation or abnormal coagulation function in the past;
5. Clinical trial participants who have previously participated in the treatment of flumiphene;
6. Other situations where the researcher deems it inappropriate to participate in the study.

Ages: 5 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Times of pulmonary hemorrhage | 12 months
  Annual times of acute episodes of pulmonary hemorrhage

SECONDARY OUTCOMES:
Rate of adverse reaction | 12 months
  The frequency of adverse reactions and their relationship with leflunomide

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China